CLINICAL TRIAL: NCT05351918
Title: Migraine Treatment With Acupuncture: Comparison of Standard Protocol to Meridian Based Protocol
Brief Title: Comparison of Two Different Migraine Acupuncture Treatment
Status: Completed | Type: Observational
Sponsor: University Medical Centre Ljubljana (Other)
Responsible Party: Principal Investigator, Jasmina Markovic Bozic, asist. prof., PhD, University Medical Centre Ljubljana
Other Study IDs: 0120-434/2021/7
Record Dates: First submitted 2022-04-15; First posted 2022-04-28 (Actual); Last update posted 2022-11-09 (Actual); Status verified 2022-11

CONDITIONS: Migraine
MeSH Terms: conditions — Migraine Disorders | interventions — Acupuncture Therapy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- migrain days: Two methods of acupuncture stimulation will be compared. In all patients, DU 20 point and the same distal points will be used.
  In the control group, all patients will receive the same local points, commonly used to treat migraine in our department.
  In the study group, local points will be selected according to the site of the headache.
  Interventions: Other: acupuncture
- consumption of analgesics: Two methods of acupuncture stimulation will be compared. In all patients, DU 20 point and the same distal points will be used.
  In the control group, all patients will receive the same local points, commonly used to treat migraine in our department.
  In the study group, local points will be selected according to the site of the headache.
  Interventions: Other: acupuncture

INTERVENTIONS:
Other: acupuncture — Acupuncture points are punctured with needles.

SUMMARY:
Headache is one of the most common clinical problems. Conventional drug therapy is more successful when complementary and integrative medicine approaches are combined to conventional treatment, as traditional Chinese medicine (TKM).

The success of acupuncture therapy depends on the selection of acupuncture points according to TKM pathological mechanisms. Correct selection of points are needed to treat migraine headaches.Acupuncture reduces the consumption of analgesics.

In this prospective, randomised study we will compered two methods of acupuncture stimulation: in the control group, all patients will receive the same local points, commonly used to treat migraine in our department, in the study group, local points will be selected according to the site of the headache.

DETAILED DESCRIPTION:
Headache is one of the most common clinical problems. It is a subjective symptom that can be associated with many other syndromes. Conventional drug therapy is often effective in reducing of acute headache and also in the frequency and intensity of chronic headaches. However, the treatment is even more successful when complementary and integrative medicine approaches are combined to conventional treatment. The most commonly used method is traditional Chinese medicine (TKM).

Although acupuncture has been a key component of TKM for more than 2500 years, the mechanism of action is still not fully understood. Acupuncture needles probably stimulates the delta fibers, and thus the pain stimulus does not occur to the talamus. Acupuncture increases the activity of the opioidergic system by releasing serotonin, dopamine, neurotrophines and nitric oxide, which are effective in treating chronic pain and migraines. Acupuncture has been recognised by the WHO as a method for the treatment of acute and chronic pain. The success of acupuncture therapy depends on the selection of acupuncture points according to TKM pathological mechanisms. Correct selection of points are needed to treat migraine headaches. Local, regional and distal points are used. Acupuncture reduces the consumption of analgesics.

The research will be conducted in the clinical Department of Anaesthesiology and Intensive Care Therapy in University Medical Centre Ljubljana. Patients with migraine headaches will be included in the study. The quality of life after treatment, drug consumption, satisfaction and well-being will be monitored. The research will determine if targeted acupuncture stimulation regard to the location of headache reduces the frequency and severity of migraines compared to the established treatment method, thus reducing the number diabled days. The added value of the research is monitoring the quality of life after completed treatment, drug consumption and in satisfaction and well-being of the patient.

PROTOCOL

60 patients with migraine will be included in this prospective, randomised study, scheduled for acupuncture stimulation. Two methods of acupuncture stimulation will be compared. In all patients, DU 20 point and the same distal points will be used.

• ALL PATIENTS: DU 20 local points: Ex 1 distal points: LI 4, St 36, Liv 2

In the control group, all patients will receive the same local points, commonly used to treat migraine in our department.

• CONTROL GROUP: localn points: UB 2; GB 14, 16, 20 distal points: PC 6, SJ 5

In the study group, local points will be selected according to the site of the headache.

ELIGIBILITY:
Inclusion Criteria:

* age >18 years
* pragnancy

Exclusion Criteria:

* patients refusal

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with migrain
Sampling Method: Probability Sample
Enrollment: 48 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2022-04-15 (Actual); Study Completion 2022-04-15 (Actual)

PRIMARY OUTCOMES:
number disabled migraine days | 6 months
  The quality of life after treatment, drug consumption, satisfaction and well-being will be monitored. The research will determine if targeted acupuncture stimulation regard to the location of headache reduces the frequency and severity of migraines compared to the established treatment method, thus reducing the number diabled days. The added value of the research is monitoring the quality of life after completed treatment, drug consumption and in satisfaction and well-being of the patient.

CONTACTS AND LOCATIONS:
Overall Officials: Jasmina Markovic - Bozic, PhD, Principal Investigator — UMC LJUBLJANA
Locations (1):
- UMC Ljubljana, Ljubljana, Slovenia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] 1. Headache Classification Committee of the International Headache Society (IHS) The International Classification of Headache Disorders, 3rd edition. Cephalalgia. 2018 Jan;38(1):1-211. 2. Goadsby PJ. Pathophysiology of migraine. Neurol Clin. 2009 May;27(2):335-60. 3. Zobdeh F, Kraiem AB, Attwood MM, et al. Pharmacological treatment of migraine: Drug classes, mechanisms of action, clinical trials and new treatments. Br J Pharmacol. 2021 Dec;178(23):4588-4607. 4. Millstine D, Chen CY, Bauer B. Complementary and integrative medicine in the management of headache. BMJ. 2017 May 16;357:j1805. 5. Rajapakse T, Pringsheim T. Nutraceuticals in Migraine: A Summary of Existing Guidelines for Use. Headache. 2016 Apr;56(4):808-16. 6. Rožman P, Osojnik J. Tradicionalna kitajska medicina in akupunktura, 1.del. Slovensko društvo za orientalno medicino. Ljubljana. 1993. 7. Lozano F. Pattern Discrimination in Traditional Chinese Medicine (TCM). In: Lin YC, Hsu EZ, eds. Acupuncture for Pain Management. New York: Springer; 2014. p. 45-72 8. Zhao L, Chen J, Li Y, et al. The Long-term Effect of Acupuncture for Migraine Prophylaxis: A Randomized Clinical Trial. JAMA Intern Med. 2017 Apr 1;177(4):508-515. 9. Liu Y, Yu S. Recent Approaches and Development of Acupuncture on Chronic Daily Headache. Curr Pain Headache Rep. 2016 Jan;20(1):4. 10. Langevin HM, Bouffard NA, Badger GJ, et al. Subcutaneous tissue fibroblast cytoskeletal remodeling induced by acupuncture: evidence for a mechanotransduction-based mechanism. J Cell Physiol. 2006 Jun;207(3):767-74. 11. Keown D. The spark in the machine. London and Philadelphia: Singing Dragon; 2014. 12. Hwang YC, Lee IS, Ryu Y, et al. Exploring traditional acupuncture point selection patterns for pain control: data mining of randomised controlled clinical trials. Acupunct Med. 2020 Jun 20 13. Silva Andrade B, Siqueira S, de Assis Soares WR, et al. Long-COVID and Post-COVID Health Complications: An Up-to-Date Review on Clinical Conditions and Their Possible Molecular Mechanisms. Viruses. 2021 Apr 18;13(4):700. 14. Martelletti P, Bentivegna E, Spuntarelli V, et al. Long-COVID Headache. SN Compr Clin Med. 2021;3(8):1704-1706.